CLINICAL TRIAL: NCT04147364
Title: Patterns of Injury and Mortality in Free-fall Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201909071RINB
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2019-10

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — only retrospective reviews for medical records

SUMMARY:
In this study, the investigator aimed to analyze the demographic characteristics, patterns of injury and mortality after free fall in a Taiwan level one trauma center.

DETAILED DESCRIPTION:
Falls from height is the leading cause of accidental deaths. The mechanism of free-fall injury is abrupt vertical deceleration and the severity is dependent on the height, body weight, posture and contact area…etc. Most victims presented to emergency department with major trauma, so initial evaluation and timely management are crucial for the survival. The knowledge of unique pattern of injuries helps clinicians to facilitate the diagnosis. In this study, the investigator aimed to analyze the demographic characteristics, patterns of injury and mortality after free fall in a Taiwan level one trauma center.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with free-fall trauma

Exclusion Criteria:

* adult patients with free-fall trauma, not relating with traffic accidents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patterns of injury and mortality after free-falls in a Taiwan level one trauma center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
patterns of injury and causes of mortality | one month
  patterns of injury and causes of mortality in free-fall patients

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Emergency Department, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No